CLINICAL TRIAL: NCT00827099
Title: Transplantation of Two Partially Matched Umbilical Cord Blood Units Following Reduced Intensity Conditioning to Enhance Engraftment and Limit Transplant-Related Mortality in Adults With Hematologic Malignancies
Brief Title: Umbilical Cord Blood (UCB) Transplant, Fludarabine, Melphalan, and Anti-thymocyte Globulin (ATG) in Treating Patients With Hematologic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unacceptable morbidity & mortality
Sponsor: Northside Hospital, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000632453; BMTGG-NSH-801
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Results first posted 2011-08-03 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: accelerated phase cml; adult ALL in remission; adult AML in remission; adult AML with 11q23 (MLL) abnormalities; adult AML with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); blastic phase chronic myelogenous leukemia; chronic myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; prolymphocytic leukemia; recurrent adult T-cell leukemia/lymphoma; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; refractory chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent adult Hodgkin lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; cutaneous B-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; adult grade III lymphomatoid granulomatosis; adult nasal type extranodal NK/T-cell lymphoma; Waldenstrom macroglobulinemia; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult grade III lymphomatoid granulomatosis; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; chronic idiopathic myelofibrosis; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Prolymphocytic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Lymphoma, Extranodal NK-T-Cell; Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Primary Myelofibrosis | interventions — Antilymphocyte Serum; fludarabine phosphate; Melphalan; Mycophenolic Acid; Tacrolimus; Cord Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: anti-thymocyte globulin — anti-thymocyte globulin
Drug: fludarabine phosphate — fludarabine phosphate
Drug: Melphalan — melphalan
Drug: mycophenolate mofetil — mycophenolate mofetil
Drug: tacrolimus — tacrolimus
Procedure: umbilical cord blood transplantation — umbilical cord blood transplantation

SUMMARY:
RATIONALE: Giving low doses of chemotherapy before a donor umbilical cord blood transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving tacrolimus and mycophenolate mofetil after the transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well giving umbilical cord blood transplant together with fludarabine, melphalan, and antithymocyte globulin works in treating patients with hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the 100-day transplant-related (non-relapse) mortality in patients with hematologic malignancies undergoing reduced-intensity conditioning comprising fludarabine phosphate, melphalan, and anti-thymocyte globulin followed by sequential umbilical cord blood transplantation (UCBT) from 2 partially-matched unrelated donors.

Secondary

* To evaluate the 12-month transplant-related (non-relapse) mortality.
* To evaluate the days to neutrophil engraftment (ANC > 500/mm³).
* To evaluate the days to platelet engraftment (platelet count > 20,000/mm³ [unsupported]).
* To evaluate the risk of acute and chronic graft-vs-host disease.
* To evaluate percent donor chimerism contribution of each cord unit.
* To evaluate relapse rate.
* To evaluate disease-free and overall survival.
* To evaluate transfusion support needed for UCBT recipients.

OUTLINE:

* Conditioning regimen: Patients receive fludarabine phosphate IV over 30 minutes on days -7 to -3, melphalan IV over 30-60 minutes on day -2, and anti-thymocyte globulin IV over 4-6 hours on days -4 to -2.
* Transplantation: Patients undergo two sequential umbilical cord blood transplantations on day 0.
* Graft-vs-host disease (GVHD) prophylaxis: Patients receive tacrolimus IV continuously and then orally twice daily beginning on day -1 and continuing until day 60, followed by a taper until day 180 in the absence of GVHD. Patients also receive mycophenolate mofetil IV or orally twice daily beginning on day 0 and continuing until day 30, followed by a taper until day 60 in the absence of GVHD.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of hematologic malignancy for which a reduced-intensity allogeneic stem cell transplantation is deemed clinically appropriate, including any of the following:

  * Chronic myelogenous leukemia, meeting one of the following criteria:

    * In first chronic phase AND failed imatinib mesylate therapy, defined as failure to obtain a hematologic remission by 3 months or major cytogenetic response (Ph+ cells < 35%) by 12 months, or demonstrated clonal evolution or disease progression while on therapy
    * In accelerated phase with < 15% blasts
    * In blast crisis that has entered into a second chronic phase following induction chemotherapy
  * Acute myelogenous leukemia, meeting one of the following criteria:

    * In second or subsequent completion remission*
    * Failed primary induction chemotherapy, but subsequently entered into a complete remission* with ≤ 2 subsequent re-induction chemotherapy treatment(s)
    * In first complete remission* with poor-risk cytogenetics NOTE: *Complete remission is defined as < 5% blasts in bone marrow, no definitive evidence of disease by morphology, flow cytometry, or genetic studies, and no circulating blasts. Neutrophil and platelet count recovery will not be required.
  * Acute lymphoblastic leukemia, meeting one of the following criteria:

    * In second or subsequent complete remission
    * In first complete remission AND t(9;22)
  * Myelodysplastic syndromes, meeting the following criteria:

    * High-risk disease, defined as International Prognostic Scoring System score of ≥ 1.5
    * Less than 10% blasts at the time of study enrollment
  * Chronic myelomonocytic leukemia

    * Less than 10% blasts at the time of study enrollment
  * Myeloid metaplasia with myelofibrosis with poor-risk features, meeting one of the following criteria:

    * Age < 55 years AND a Lille score of 1
    * Lille score of 2
    * Hemoglobin < 10 g/dL AND abnormal karyotype
  * Chronic lymphocytic leukemia/prolymphocytic leukemia, meeting all of the following criteria:

    * Rai stage I-IV disease
    * Failed ≥ 1 prior chemotherapy regimen, including fludarabine, or autologous stem cell transplantation
    * Chemosensitive or stable, non-bulky disease prior to transplant
    * Received ≤ 3 prior chemotherapy regimens (monoclonal antibody therapy and involved-field radiotherapy are not considered prior regimens)
  * Low-grade B-cell non-Hodgkin lymphoma (NHL) (small lymphocytic lymphoma, follicular center [grade 1 or 2] lymphoma, or marginal zone lymphoma), meeting all of the following criteria:

    * Failed ≥ 1 prior chemotherapy regimen or autologous stem cell transplantation
    * Chemosensitive or stable, non-bulky disease prior to transplant
    * Received ≤ 3 prior chemotherapy regimens (monoclonal antibody therapy and involved-field radiotherapy are not considered prior regimens)
  * Intermediate-grade B-cell or T-cell NHL or mantle cell NHL, meeting all of the following criteria:

    * Failed to achieve remission or recurred after either conventional chemotherapy or autologous stem cell transplantation
    * Chemosensitive, non-bulky disease prior to transplant
  * Hodgkin lymphoma, meeting all of the following criteria:

    * Relapsed after prior autologous stem cell transplantation or after ≥ 2 combination chemotherapy regimens AND ineligible for autologous peripheral blood stem cell transplantation
    * Chemosensitive, non-bulky disease prior to transplant
  * Multiple myeloma, meeting one of the following criteria:

    * Relapsed after autologous stem cell transplantation
    * Relapsed after conventional therapies AND not a candidate for autologous stem cell transplantation
* No HLA-matched related or unrelated donor available
* Has two umbilical cord blood units available that are matched at ≥ 4/6 HLA A, B, and DRB1 with the patient and with each other (HLA C and DQ will not be used in the match strategy)

  * Total combined nucleated cell dose from the 2 umbilical cord blood units must be > 3.7 x 10^7 nucleated cells/kg (pre-freeze dose) NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

* Karnofsky performance status 80-100%
* Adapted, weighted Charlson Comorbidity Index < 3
* Serum creatinine ≤ 2.0 mg/dL
* AST or ALT < 3 times upper limit of normal (ULN)
* Bilirubin < 1.5 times ULN
* Not pregnant or nursing
* LVEF ≥ 40%
* DLCO > 50%
* No hypoxia at rest with oxygen saturation < 92% on room air (corrected with bronchodilator therapy)
* No active opportunistic infection (e.g., fungal pneumonia, tuberculosis, or viral infection)
* No active hepatitis B or C infection that, in the opinion of a gastroenterologist or the transplant committee, places the patient at moderate- to high-risk for developing severe hepatic disease
* No HIV infection

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott R. Solomon, MD, Principal Investigator — Blood and Marrow Transplant Group of Georgia
Locations (1):
- Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was IRB approved on 6/8/06. The first patient was enrolled on 6/9/06. The last patient was enrolled on 12/22/08.
Pre-assignment Details: There were no group assignments for this study. It was a single arm cord blood transplant study.
Groups:
- Umbilical Cord Blood Transplantation: 1. Fludarabine 30 mg^m2 on days -7, -6, -5, -4 & -3
  2. Melphalan 140 mg^m2 on day -2
  3. Rabbit antithymocyte globulin (ATG) 6mg/kg divided over 3 days, Days -4,-3,-2. (Thymoglobulin 1.0mg/kg on day -4, and 2.5mg/kg/d on days -3, -2)
  4. Tacrolimus starting on day -1 as a continuous infusion of 0.03 mg/kg/d.
  5. Mycophenolate mofetil (MMF) IV 15mg/kg BID will start on Day 0
Period: Overall Study
Arm/Group | Umbilical Cord Blood Transplantation
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Umbilical Cord Blood Transplantation
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 35.8 (9.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 100 Day Transplant-related Mortality (TRM)
Description: 100 Day TRM is death within 100 days from transplant related complications
Time Frame: 100 days
Measure: Number; unit: participants
Groups:
- Umbilical Cord Blood Transplant: High dose conditioning with Fludarabine & Melphalan
Arm/Group | Umbilical Cord Blood Transplant
Number analyzed (Participants) | 5
participants | 0

2. Secondary Outcome: Number of Patients That Engrafted Blood Counts by 30 Days After Transplant
Description: Number of patients whose Absolute Neutrophil Count (ANC) recovered to >500 x10^3/uL for at least 3 consecutive days after transplant
Time Frame: Day 30
Measure: Number; unit: participants
Arm/Group | Umbilical Cord Blood Transplant
Number analyzed (Participants) | 5
participants | 5

3. Secondary Outcome: Percentage of Donor and Host Chimerism of Each Cord Blood Unit
Description: Evaluate the percentages of donor and host chimerism at multiple times post-transplant including Day 30, Day 60, Day 90 and monthly thereafter if the patient is not considered to have full chimerism.
Time Frame: day 30, day 60, day 90
Population: This study was terminated early. No participants were analyzed.
Measure: Number; unit: percentage of chimerism
Arm/Group | Umbilical Cord Blood Transplant
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Patients Who Experience Acute and Chronic Graft-vs-host Disease After Transplant.
Description: Patients will be evaluated regularly for the development of graft versus host disease both acute & chronic.
Time Frame: Day 30
Population: This study was terminated early. No participants were analyzed.
Measure: Number; unit: participants
Arm/Group | Umbilical Cord Blood Transplant
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Patients Who Experience Disease Relapse Post-transplant
Description: Patients will have routine restaging to assess disease response at Day 100, 6 months, 1 year, 18 months and 24 months. If disease relapse is suspected, the patient will be evaluated at that time.
Time Frame: Day 100, 6 months, 1 year, 18 months, 24 months
Population: This study was terminated early. No participants were analyzed.
Measure: Number; unit: participants
Arm/Group | Umbilical Cord Blood Transplant
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Patients Who Survive Following Treatment on This Protocol
Description: Patients will be followed until death
Time Frame: Through Death
Population: This study was terminated early. No participants were analyzed.
Measure: Number; unit: participants
Arm/Group | Umbilical Cord Blood Transplant
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Umbilical Cord Blood Transplantation
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Umbilical Cord Blood Transplantation (N=5)
Anorexia (Gastrointestinal disorders) | 4 (4)
Cognitive Disturbance - unable to verbalize (Nervous system disorders) | 2 (2)
Cognitive disturbance - incomprehensible speech (Nervous system disorders) | 2 (2)
Confusion (Nervous system disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Constitutional Symptoms - weakness (General disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Decreased Hemoglobin (Blood and lymphatic system disorders) | 4 (4)
Decreased Leukocytes (total WBC) (Blood and lymphatic system disorders) | 4 (4)
Decreased Neutrophils/Granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 4 (4)
Dehydration (Gastrointestinal disorders) | 1 (1)
Dermatology/Skin - Nail slough (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatology/Skin - nail burning (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatology/Skin - skin sensitivity (Skin and subcutaneous tissue disorders) | 2 (2) — including soles of feet
Dermatology/skin - "cut on skin" (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatology/skin - clubbing of fingernails (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatology/skin - discoloration of fingernails (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatology/skin - irritation (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatology/skin- burning palms (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema (Musculoskeletal and connective tissue disorders) | 1 (1)
Elevated ALK PHOS (Metabolism and nutrition disorders) | 1 (1)
Elevated ALT (Hepatobiliary disorders) | 2 (2)
Elevated AST (Blood and lymphatic system disorders) | 2 (2)
Elevated PTT (Metabolism and nutrition disorders) | 1 (1)
Elevated creatinine (Renal and urinary disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 1 (1)
Extremity - lower (unsteady gait) (Musculoskeletal and connective tissue disorders) | 1 (1)
Fatigue (General disorders) | 4 (4) — fatigue & drowsiness
Fever (General disorders) | 5 (5)
Flushing (Skin and subcutaneous tissue disorders) | 2 (2)
Gastrointestinal - abdominal tenderness (Gastrointestinal disorders) | 2 (2)
Gastrointestinal - tickle in throat (Gastrointestinal disorders) | 1 (1)
Gastrointestinal-other (early satiety) (Gastrointestinal disorders) | 1 (1)
Heartburn/dyspepsia (Gastrointestinal disorders) | 2 (2)
Hemorrhage - GU (hemorrhagic cystitis) (Renal and urinary disorders) | 1 (1)
Hemorrhage - GU (vaginal bleeding) (Reproductive system and breast disorders) | 1 (1)
Hemorrhage - oral cavity (Gastrointestinal disorders) | 1 (1)
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Cardiac disorders) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 5 (5)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Hypotension (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection - general bacteria (Infections and infestations) | 1 (1)
Infection - BK virus (Infections and infestations) | 2 (2)
Infection - CMV (Infections and infestations) | 3 (3)
Infection - Clostridium Difficile (Infections and infestations) | 1 (1)
Infection - HHV6 (Infections and infestations) | 1 (1)
Infection - MRSA (Infections and infestations) | 1 (1)
Infection - MRSE (Infections and infestations) | 1 (1)
Infection - corynebacterium (Infections and infestations) | 1 (1)
Infection - enterococcus faecium (Infections and infestations) | 1 (1)
Infection - pneumonia (Infections and infestations) | 1 (1)
Infection - strep mitis (Infections and infestations) | 1 (1)
Infection - strep viridans (Infections and infestations) | 1 (1)
Infection - thrush (Infections and infestations) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Lymphatics - spongiosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Memory impairment - short attention span (Nervous system disorders) | 1 (1)
Memory impairment - short term memory loss (Nervous system disorders) | 1 (1)
Mood alteration - aggitated/restless (Nervous system disorders) | 3 (3)
Mood alteration - anxiety (Nervous system disorders) | 2 (2)
Mood alteration - depression (Nervous system disorders) | 2 (2)
Mood alteration - flat affect (Nervous system disorders) | 1 (1)
Mood alteration - tearful (Nervous system disorders) | 2 (2)
Mood alteration - withdrawn (Nervous system disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 4 (4)
Musculoskeletal/Soft Tissue - Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal/soft tissue - aching in legs (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal/soft tissue - arhthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 5 (5)
Neurology (hallucinations) (Psychiatric disorders) | 1 (1)
Neuropathy - sensory (peripheral neuropathy) (Nervous system disorders) | 1 (1)
Ocular/Visual - Itching eyes (Eye disorders) | 1 (1)
Ocular/Visual - tearing eyes (Eye disorders) | 1 (1)
Ocular/visual - dilated pupils (Eye disorders) | 1 (1)
Ocular/visual - stinging eyes (Eye disorders) | 2 (2)
Pain - Cardiovascular (chest pain) (Cardiac disorders) | 1 (1)
Pain - Gastrointestinal (throat pain) (Gastrointestinal disorders) | 2 (2)
Pain - General (pain NOS) (General disorders) | 3 (3)
Pain - Neurology (headache) (General disorders) | 5 (5)
Pain - musculoskeletal (back pain) (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - sexual/reproductive function (vaginal pain) (Reproductive system and breast disorders) | 1 (1)
Pruritis/itching (Skin and subcutaneous tissue disorders) | 4 (4)
Pulmonary/Upper Respiratory - Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/Upper Respiratory - sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Renal/Genitourinary - difficulty urinating (Renal and urinary disorders) | 1 (1)
Renal/Genitourinary - dysuria (Renal and urinary disorders) | 3 (3)
Renal/Genitourinary - prostate enlargement (Renal and urinary disorders) | 1 (1)
Renal/Genitourinary - sphincter spasms (Renal and urinary disorders) | 1 (1)
Renal/Genitourinary - urinary hesitancy (Renal and urinary disorders) | 1 (1)
Rigors/chills (General disorders) | 4 (4)
Seizure (Nervous system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
Tremor (Nervous system disorders) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 2 (2)
Ventricular arrhythmia - tachycardia (Cardiac disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Watery eye (Eye disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated early, therefore no additional data measures or outcomes are available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No